CLINICAL TRIAL: NCT00859586
Title: Mismatched Donor Lymphocyte Infusions for Relapsed Disease Following Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090087; 09-H-0087 (Other: NIH NHLBI)
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2014-08

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphoblastic, Acute; Leukemia, Myelocytic, Chronic
Keywords: Acute Myelogenous Leukemia (AML); Acute Lymphoblastic Leukemia (ALL); Chronic Lymphocytic Leukemia; Myelodysplastic Syndrome (MDS); Acute Myelogenous Leukemia; AML; Acute Lymphoblastic Leukemia; ALL; Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: The CliniMACS CD34 Reagent System is a medical device used in vitro to select and enrich specific cell populations (CD34+ cells from heterogeneous hematological cell populations). In stage 1, subjects will receive 1 x 108 CD3 cells/kg on day 0. We will progress to stage 2 where the dose of CD3+ cells will be increased to 2 x 108 cells/kg.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Miltenyi Magnetic cell sorter for CD3 (Experimental): Miltenyi Magnetic cell sorter device will be used for CD3 selection of granulocyte colony stimulating factor mobilized allogeneic PBSCT. In stage 1, subjects will receive 1 x 10 to the eight power CD3 cells/kg. In stage II, the dose of CD3+ cells will be increased to 2 x 10 to the eight power cells/kg.
  This phase II clinical trial is designed to evaluate a novel non-myeloablative but highly immunosuppressive disease specific conditioning regimen and infusion of unmanipulated lymphocytes from a haplo-identical familial donor in subjects with relapsed disease following matched sibling stem cell transplantation who are not candidates for alternative treatment options. The clinical trial will evaluate recipient survival at six months post-relapse of disease.
  Interventions: Device: Miltenyi Magnetic cell sorter for CD3

INTERVENTIONS:
Device: Miltenyi Magnetic cell sorter for CD3 — Receipts will receive 1 x 10 to eighth power CD3 cells/kg of familial haploidentical positively selected cluster of differentiation 34 (CD34)+ stem cells from the same DLI donor.
  Other Names: CliniMACS Miltenyi

SUMMARY:
Patients receiving allogeneic stem cell transplantation for hematological malignancies who suffer a relapse of their disease post-transplant have limited treatment options and a poor prognosis. With the exception of patients with chronic leukemias who may achieve prolonged remissions after donor lymphocyte infusions (DLIs), treatments using either chemotherapy or a DLI achieve less than a 10% median survival beyond 6 months. Most of these patients die of progressive leukemia, underlying the need for new therapeutic approaches.

Human leukocyte antigen (HLA)-mismatched DLIs appear to possess a more potent graft-versus-leukemia (GvL) effect. However, when given after an HLA-mismatched transplant DLIs have a high risk of causing graft-versus-host disease (GvHD), which can be severe. To reduce the risk of GvHD, infusions of mismatched lymphocytes from an alternative donor may be used to avoid permanent engraftment and associated risk of GvHD.

In this study, we propose to use a novel strategy to treat leukemias relapsing after HLA matched allogeneic stem cell transplantation by using haplo-identical DLIs to promote the associated antileukemic effect while minimizing the possibility of permanent engraftment and associated GvHD. To achieve only temporary engraftment and to promote disease control we will give fludarabine immunosuppression prior to the DLI. We anticipate the infusion of HLA-mismatched donor lymphocytes in this setting will produce no detectible engraftment or only temporary engraftment, but may result in a strong GvL effect regardless of engraftment outcome. We will select patients for this protocol who fall into the worst category for post-transplant relapse. Specifically, we will enroll patients with acute leukemia or MDS relapsing within 6 months of transplant, of which less than 5% survive beyond a year from relapse.

DETAILED DESCRIPTION:
Patients receiving allogeneic stem cell transplantation for hematological malignancies who suffer a relapse of their disease post-transplant have limited treatment options and a poor prognosis. With the exception of patients with chronic leukemias who may achieve prolonged remissions after donor lymphocyte infusions (DLIs), treatments using either chemotherapy or a DLI achieve less than a 10% median survival beyond 6 months. Most of these patients die of progressive leukemia, underlying the need for new therapeutic approaches.

HLA-mismatched DLIs appear to possess a more potent graft-versus-leukemia (GvL) effect. However, when given after an HLA-mismatched transplant DLIs have a high risk of causing graft-versus-host disease (GvHD), which can be severe. To reduce the risk of GvHD, infusions of mismatched lymphocytes from an alternative donor may be used to avoid permanent engraftment and associated risk of GvHD.

In this study, we propose to use a novel strategy to treat leukemias relapsing after HLA matched allogeneic stem cell transplantation by using haplo-identical DLIs to promote the associated antileukemic effect while minimizing the possibility of permanent engraftment and associated GvHD. To achieve only temporary engraftment and to promote disease control we will give fludarabine immunosuppression prior to the DLI. We anticipate the infusion of HLA-mismatched donor lymphocytes in this setting will produce no detectible engraftment or only temporary engraftment, but may result in a strong GvL effect regardless of engraftment outcome. We will select patients for this protocol who fall into the worst category for post-transplant relapse. Specifically, we will enroll patients with acute leukemia or MDS relapsing within 6 months of transplant, of which less than 5% survive beyond a year from relapse.

The primary objective of this phase II clinical trial will be to evaluate the safety and efficacy of using a non-engraftment model and a lymphocytes infusion from a haplo-identical donor to treat relapsed disease following matched sibling stem cell transplantation in subjects who are not candidates for alternative treatment options.

We therefore propose this is a phase II clinical trial is to evaluate the safety and efficacy of an infusion of unmanipulated lymphocytes from a haplo-identical donor in subjects with relapsed disease following matched sibling stem cell transplantation who are not candidates for alternative treatment options.

The primary endpoint of this phase 2 study is survival at 6 month post-relapse of disease. Successful outcome of the study will be a survival of 100% greater than the National Heart Lung and Blood (NHLBI) historical 25% at 6-months.

Secondary endpoints will include: incidence and severity of induced GvHD, proportion of DLI engraftment, peak chimerism, leukemia response at 21 days post DLI, residual leukemia measured by patient chimerism, leukemia free survival from date relapse, and safety of the mismatched DLI procedure.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Inclusion Criteria- Recipient:

1. Diagnosed with one of the following hematological conditions:

   * Acute lymphoblastic leukemia (ALL) of any subtype or
   * Acute myelogenous leukemia (AML) of any subtype or
   * Myelodysplastic syndrome (MDS) of any subtype or
   * Blastic phase Chronic Myeloid Leukemia (CML)
2. Relapsed disease within 6 months of matched sibling allogeneic stem cell transplant procedure
3. Evaluation for protocol within 8 weeks of relapse and enrollment within 12 weeks or relapse
4. 8-75 years of age
5. Availability of previous HLA identical (6/6) related donor (ages 8 to 17 must have previously donated bone marrow [not peripheral blood]
6. At least one haploidentical (1-3 antigen mismatched) related donor available for apheresis

Exclusion Criteria Recipient (any of the following):

1. Active grade II-IV Graft vs. Host Disease (GvHD)
2. Extensive chronic Graft vs. Host Disease (GvHD)
3. Post-transplant donor lymphocyte infusion (DLI) from original donor within 1 month of protocol enrollment.
4. Progressive disease despite post-relapse chemo or monoclonal therapy.
5. Co-morbidity of such severity that it would preclude the patients ability to tolerate protocol therapy.
6. Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) greater than 10 x ULN (grade 3, CTCAE).
7. Bilirubin greater than 5 x Upper Limit of Normal (ULN) (grade 3, CTCAE).
8. Creatinine greater than 3.5 mg/dl (grade 3, CTCAE).
9. HIV positive (Recipients who are positive for hepatitis B (HBV), hepatitis C (HCV) or human T-cell lymphotropic virus (HTLV-I/II) are not excluded from participation).
10. Positive pregnancy test for women of childbearing age.
11. Severe psychiatric illness or mental deficiency sufficiently severe as to make compliance with the transplant treatment unlikely and informed consent impossible.

Inclusion Criteria- Stem Cell Donors:

1. HLA-matched sibling stem cell donor from the original transplant to participate in a stem cell rescue only in the setting of severe, refractory GvHD caused by the haploidentical cells.
2. Related HLA haplo-identical (1-3 A, B or DR antigens mismatched with recipient). To maximize the GvL that is associated with HLA disparity, the haploidentical donor will be chosen based on the greatest HLA mismatch (preference: 3/6 greater than 4/6 greater than 5/6). Parents and siblings will be considered equally.
3. Weight greater than or equal to 18 kg
4. Age greater than or equal to 8 or less than or equal to 80 years old.

Exclusion Criteria Stem Cell Donor (any of the following):

1. Pregnant or lactating
2. Unfit to receive filgrastim (G-CSF) or previous filgrastim mobilization for donors under 18 years of age.
3. Unfit to undergo apheresis (abnormal blood counts, history of stroke, uncontrolled hypertension).
4. Sickling hemoglobinopathies such as HbSS or HbSC.
5. HIV positive. Donors who are positive for hepatitis B (HBV), hepatitis C (HCV), human T-cell lymphotropic virus (HTLV-I/II), or T.cruzi (Chagas) will be used at the discretion of the investigator following counseling and approval from the recipient.
6. Severe psychiatric illness or mental deficiency sufficiently severe as to make compliance with the donation of stem cells unlikely and/or informed consent impossible.

Inclusion criteria- Haplo Lymphocyte Donors:

1. Related HLA haplo-identical (1-3 A, B or DR antigens mismatched with recipient). To maximize the GvL that is associated with HLA disparity, the haploidentical donor will be chosen based on the greatest HLA mismatch (preference: 3/6 greater than 4/6 greater than 5/6). Donors age less than 80 years required, and parents and siblings will be considered equally.
2. Age greater than or equal to 18 or less than or equal to 80 years old.

Exclusion Criteria Haplo Lymphocyte Donor (any of the following):

1. Pregnant or lactating
2. Unfit to undergo apheresis (abnormal blood counts, history of stroke, uncontrolled hypertension).
3. Sickling hemoglobinopathies such as HbSS and HbSC .
4. HIV positive. Donors who are positive for hepatitis B (HBV), hepatitis C (HCV) or human T-cell lymphotropic virus (HTLV-I/II), or T.cruzi (Chagas) will be used at the discretion of the investigator following counseling and approval from the recipient.
5. Severe psychiatric illness or mental deficiency sufficiently severe as to make compliance with the donation of stem cells unlikely and/or informed consent impossible

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minoo Battiwalla, Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health, Bethesda, Maryland, United States

REFERENCES:
- [Background] Armitage JO. Bone marrow transplantation. N Engl J Med. 1994 Mar 24;330(12):827-38. doi: 10.1056/NEJM199403243301206. No abstract available. PMID 8114836
- [Background] Montero A, Savani BN, Shenoy A, Read EJ, Carter CS, Leitman SF, Mielke S, Rezvani K, Childs R, Barrett AJ. T-cell depleted peripheral blood stem cell allotransplantation with T-cell add-back for patients with hematological malignancies: effect of chronic GVHD on outcome. Biol Blood Marrow Transplant. 2006 Dec;12(12):1318-25. doi: 10.1016/j.bbmt.2006.08.034. PMID 17162214
- [Background] Levine JE, Braun T, Penza SL, Beatty P, Cornetta K, Martino R, Drobyski WR, Barrett AJ, Porter DL, Giralt S, Leis J, Holmes HE, Johnson M, Horowitz M, Collins RH Jr. Prospective trial of chemotherapy and donor leukocyte infusions for relapse of advanced myeloid malignancies after allogeneic stem-cell transplantation. J Clin Oncol. 2002 Jan 15;20(2):405-12. doi: 10.1200/JCO.2002.20.2.405. PMID 11786567
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-H-0087.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Started | 8
Completed | 4
Not Completed | 4
Not completed — Donors | 4

BASELINE CHARACTERISTICS:
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Recipient Survival at 6-month Post-relapse of Disease
Description: This phase II clinical trial is designed to evaluate a novel non-myeloablative but highly immunosuppressive disease specific conditioning regimen and infusion of unmanipulated lymphocytes from a haplo-identical familial donor in subjects with relapsed disease following matched sibling stem cell transplantation who are not candidates for alternative treatment options. The clinical trial will evaluate recipient survival at six months post-relapse of disease.
Time Frame: 6 months post-relapse of disease
Measure: Number; unit: participants
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Number analyzed (Participants) | 4
participants
  Recipent Survival | 0
  Recipient Mortality | 4

2. Secondary Outcome: Number of Participants Who Developed of Acute GVHD
Description: Overall number incidences of participants who developed Acute Graft versus Host Disease (GVHD).
Time Frame: 6 months post disease relapse
Measure: Count of Participants; unit: Participants
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Number analyzed (Participants) | 4
Participants | 2

3. Secondary Outcome: Number of Participants Who Developed Grade I, Acute GVHD
Description: Number of participants who developed Grade I, Acute Graft vs Host Disease (GVHD) as defined by CIMBTR criteria for Organ Stages of Acute GVHD.
  Grade 1 is defined as: Skin = Maculopapular rash< 25% of body surface area (BSA); Liver = Total Bilirubin 2-3 mg/dL; Lower GI = stool output/day is 500-999 mL/day.
  Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: 6 months post disease relapse
Measure: Count of Participants; unit: Participants
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Number analyzed (Participants) | 4
Participants | 1

4. Secondary Outcome: Number of Participants Who Developed Grade II, Acute GVHD
Description: Number of participants who developed Grade II, Acute Graft vs Host Disease (GVHD) as defined by CIMBTR criteria for Organ Stages of Acute GVHD.
  Stage II Acute GVHD: Skin - rash on 25-50 percent body surface area; Liver - Total Bilirubin 3.1-6.0 mg/dL; Lower GI - Diarrhea 1001-1500 mL/day.
  Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: 6 months post disease relapse
Measure: Count of Participants; unit: Participants
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Number analyzed (Participants) | 4
Participants | 0

5. Secondary Outcome: Number of Participants Who Developed Grade III, Acute GVHD
Description: Number of participants who developed Grade III, Acute Graft vs Host Disease (GVHD) as defined by CIMBTR criteria for Organ Stages of Acute GVHD.
  Stage III Acute GVHD: Skin - Rash on >50% of body surface; Liver - Total Bilirubin 6.1 - 15.0 mg/dL; Lower GI - Diarrhea > 1500 mL/day Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: 6 months post disease relapse
Measure: Count of Participants; unit: Participants
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Number analyzed (Participants) | 4
Participants | 2

6. Secondary Outcome: Number of Participants Who Developed of Grade IV, Acute GVHD
Description: Number of participants who developed Grade IV, Acute Graft vs Host Disease (GVHD) as defined by CIMBTR criteria for Organ Stages of Acute GVHD.
  Grade IV, Acute GVHD is defined as: Skin = Generalized erythroderma plus bullous formation; Liver = Total Bilirubin >15 mg/dL; Lower GI = Severe abdominal pain with or without ileus.
  Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: 6 months post disease relapse
Measure: Count of Participants; unit: Participants
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Number analyzed (Participants) | 4
Participants | 0

7. Secondary Outcome: Number of Participants Who Developed Chronic GVHD
Description: Number of incidences of participants who developed Chronic Graft vs Host Disease (GVHD). Moderate GVHD is 3 or more organs with score 1, any organ with score 2, or lung with score 1, and usually requires systemic immune-suppressive treatment. Mild disease is associated with a good prognosis whereas severe disease is associated with higher treatment-related mortality and lower survival.
  Organs are scored on a 0 to 3 scale from no involvement/no symptoms to severe functional compromise.
Time Frame: 6 months post disease relapse
Measure: Count of Participants; unit: Participants
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Number analyzed (Participants) | 4
Participants | 0

8. Secondary Outcome: Number of Participants Who Developed Limited Chronic GVHD
Description: Number of participants who developed Limited Chronic Graft vs Host Disease (GVHD). Limited chronic GVHD is defined as GVHD occurring after day 100 that involved localized skin and/or mouth and/or liver.
Time Frame: 6 months post disease relapse
Measure: Count of Participants; unit: Participants
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Number analyzed (Participants) | 4
Participants | 0

9. Secondary Outcome: Number of Participants With Extensive, Chronic GVHD
Description: Number of participants with extensive, Chronic Graft vs Host Disease (GVHD). Extensive chronic GVHD is defined as GVHD occurring after day 100 that did not meet the definition of limited chronic GVHD.
Time Frame: 6 months post disease relapse
Measure: Count of Participants; unit: Participants
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Number analyzed (Participants) | 4
Participants | 0

10. Secondary Outcome: Number of Participants With CD3+ Engraftment Who Achieved Peak Chimerism Post DLI
Description: Number of Participants with CD3+ Engraftment who Achieved Peak Chimerism post Donor Lymphocyte Infusion (DLI)
Time Frame: 21 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Number analyzed (Participants) | 4
Participants | 3

11. Secondary Outcome: Number of Subjects Leukemia Response After Donor Lymphocyte Infusion (DLI)
Description: Subjects experience leukemia response after partially human leukocyte antigen (HLA) matched DLI according to International Working Group criteria
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: Follow up for adverse events can occur up to 6 months post disease relapse
Arm/Group | Miltenyi Magnetic Cell Sorter for CD3
All-Cause Mortality (participants affected / at risk) | 4/4
Serious Adverse Events (participants affected / at risk) | 4/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Miltenyi Magnetic Cell Sorter for CD3 (N=4)
Pulmonary Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 2 (2)
Cardiac Arrythmia (Cardiac disorders) | 1 (1)
Disease relapse (Blood and lymphatic system disorders) | 2 (2)
Multi-organ failure (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes